CLINICAL TRIAL: NCT04239755
Title: Doxycycline Effects on Neurological Outcomes in Patients With Acute Traumatic Brain Injury
Brief Title: Doxycycline in Acute Traumatic Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Clinical Pharmacy Lecturer, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Doxycycline effects on TBI
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Doxycycline; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycycline (Active Comparator): Group (1) 25 patients that receive doxycycline 100 mg twice daily, either orally or through a nasogastric tube for 5 days.
  Interventions: Drug: Doxycycline 100 MG Oral Tablet
- Placebo (Placebo Comparator): group (2) will be 25 patients will receive placebo in addition to the standard treatment.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Doxycycline 100 MG Oral Tablet — doxycycline 100 mg twice daily, either orally or through a nasogastric tube for 5 day
  Other Names: vibramycine
  Arms: Doxycycline
Other: placebo — placebo in addition to the standard treatment.
  Arms: Placebo

SUMMARY:
evaluate the impact of Doxycycline on both clinical outcome and blood levels of NSE in patients with TBI.

DETAILED DESCRIPTION:
1. Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damnhour University.
2. All Participants agreed to take part in this clinical research and provide informed consent. for unconscious participants, the informed consent was obtained from their legally authorized representative.
3. Patients with moderate to severe TBI will be enrolled from Tanta university hospitals.
4. Serum samples will be collected for measuring the biomarkers.
5. Our design is randomized, controlled study.
6. All enrolled patients will be divided into 2 groups, Group (1) 25 patients that receive doxycycline 100 mg twice daily, either orally or through a nasogastric tube for 5 days, and group (2) will be 25 patients will receive placebo in addition to the standard treatment.
7. All patients will be followed up during ICU period.
8. Statsicial tests appropriate to the study design will be conducted to evaluate the significance of the results.
9. Measuring outcome: the primary outcome is the change in the serum level of acute brain injury biomarkers.
10. Results, conclusions, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Hospital admission in the first 24 h of injury,
2. 18 to 90 years of age and
3. Both sexes with moderate to severe traumatic brain injury (GCS score ≤ 12).
4. Able to tolerate enteral feeding and drug administration within the first 24 hours of TBI

Exclusion Criteria:

1. Hypersensitivity to tetracyclines
2. Pregnant and breast feeding women,
3. History of autoimmune disease.
4. History of receiving chronic steroid treatment and isotretinoin,
5. Pre-existing hepatic (AST, ALT greater than 3 times the upper limit of normal) or renal failure (BUN/ Creatinine 20:1; creatinine > 2 mg/dL),
6. Known malignancies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Neuron specific enolase | 7 days
  levels of NSE
Glasgow Coma Scale (GCS) | 7 days
  Glasgow Coma Scale (GCS) 15 Points Normal:3 Points Abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Noha Mansour, Lecturer, Principal Investigator — Mansoura University
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sanchez Mejia RO, Ona VO, Li M, Friedlander RM. Minocycline reduces traumatic brain injury-mediated caspase-1 activation, tissue damage, and neurological dysfunction. Neurosurgery. 2001 Jun;48(6):1393-9; discussion 1399-401. doi: 10.1097/00006123-200106000-00051. PMID 11383749
- [Result] Janata A, Magnet IA, Schreiber KL, Wilson CD, Stezoski JP, Janesko-Feldman K, Kochanek PM, Drabek T. Minocycline fails to improve neurologic and histologic outcome after ventricular fibrillation cardiac arrest in rats. World J Crit Care Med. 2019 Nov 19;8(7):106-119. doi: 10.5492/wjccm.v8.i7.106. eCollection 2019 Nov 19. PMID 31853446